CLINICAL TRIAL: NCT05632029
Title: Laser Acupuncture in Systemic Lupus Women With Prediabetes
Brief Title: Laser Acupuncture in Egyptian Systemic Lupus Females With Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004113
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus; PreDiabetes
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser (active laser) (Active Comparator): 32 lupus prediabetic women will receive laser acupuncture (active laser) for one month (3 days week) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian, laser will be applied for 1 min on every acupiont)
  Interventions: Device: active laser
- laser (sham laser) (Sham Comparator): 32 lupus prediabetic women will receive laser acupuncture (sham . i.e power of the device will be zero) for one month (3 days week) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian, laser will be applied for 1 min on every acupiont)
  Interventions: Device: sham laser

INTERVENTIONS:
Device: active laser — 32 lupus prediabetic women will receive laser acupuncture (active laser) for one month (3 days week) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian, laser will be applied for 1 min on every acupiont)
  Arms: laser (active laser)
Device: sham laser — 32 lupus prediabetic women will receive laser acupuncture (sham laser, i.e power of device will be zero watt) for one month (3 days week) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian, laser will be applied for 1 min on every acupiont)
  Arms: laser (sham laser)

SUMMARY:
glucose hemosatasis, oxidative stress, abnormalities of blood pressures, and high inflammatory status is high presented in lupus patients.

DETAILED DESCRIPTION:
64 lupus prediabetic women will equally distributed to group A (n =32 that will receive laser acupuncture (active) for one month (3 days week) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian, laser will be applied for 1 min on every acupiont) or group B (n =32 this group will receive the same protocol of group A but the points will be sham points)

ELIGIBILITY:
Inclusion Criteria:

* prediabetic lupus females (n =64)

Exclusion Criteria:

* obesity diabetes heart or respiratory problems

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 64 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Malondialdehyde | It will be measured after 4 weeks of laser application
  oxidative stress indicator

SECONDARY OUTCOMES:
systolic blood pressure | It will be measured after 4 weeks of laser application
  manual sphygmomanometer
diastolic blood pressure | It will be measured after 4 weeks of laser application
  manual sphygmomanometer
blood glucose | It will be measured after 4 weeks of laser application
  it will be measured in fasting status
erythrocyte sedimentation rate (at first hour) | It will be measured after 4 weeks of laser application
  it will be measured in serum
erythrocyte sedimentation rate (at second hour) | It will be measured after 4 weeks of laser application
  it will be measured in serum
C reactive protein | It will be measured after 4 weeks of laser application
  it will be measured in serum
adenosine triphosphate | It will be measured after 4 weeks of laser application
  it a measure for energy production
Nitrate | It will be measured after 4 weeks of laser application
  it will be measured in serum
Glutathione | It will be measured after 4 weeks of laser application
  it will be measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt